CLINICAL TRIAL: NCT03429387
Title: Early Diagnosis and Treatment of Infections in Patients With Haematologic Malignancies: Examining Novel Diagnostics Including Bacterial and Fungal Multiplex PCR and FDG-PET Imaging
Brief Title: PET/CT and Bacterial/Fungal PCR in High Risk Febrile Neutropenia
Acronym: PIPPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Melbourne Health (Other); Westmead Hospital (Unknown); Victorian Infectious Diseases Reference Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/98
Record Dates: First submitted 2017-12-05; First posted 2018-02-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Haematopoietic Stem Cell Transplant, Autologous; Haematopoietic Stem Cell Transplant, Allogeneic; Febrile Neutropenia
Keywords: Diagnosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Febrile Neutropenia; Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the PET/CT arm or the conventional CT arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDG-PET/CT arm (Experimental): Participants with persistent febrile neutropenia after 72 hours of onset who are randomized to this arm will have an FDG-PET/CT performed to look for source of fever.
  Interventions: Diagnostic Test: FDG-PET/CT
- Conventional CT arm (Active Comparator): Participants with persistent febrile neutropenia after 72 hours of onset who are randomized to this arm will have a conventional CT (HRCT chest and sinuses +/- other regions as per clinician's discretion) performed to look for source of fever.
  Interventions: Diagnostic Test: Conventional CT

INTERVENTIONS:
Diagnostic Test: FDG-PET/CT — FDG-PET performed with low dose CT
  Other Names: PET/CT
  Arms: FDG-PET/CT arm
Diagnostic Test: Conventional CT — HRCT and CT of sinuses +/- other regions as per clinician's discretion
  Arms: Conventional CT arm

SUMMARY:
Patients with acute leukaemia requiring induction or consolidation chemotherapy and those requiring a haematopoietic stem cell transplant are at high risk of fever and infection when they have low white cell counts (neutropenic fever). The causes of neutropenic fever are frequently unknown and patients are treated with broad antibiotics, without a clear target to what is being treated.

This study will prospectively enroll patients who are receiving chemotherapy for acute leukaemia or for a stem cell transplant and compare the diagnostic utility of bacterial and fungal PCR performed directly off blood drawn, to the standard blood culture. Patients who have persistent fever after 72 hours of antibiotics will then be randomized to have either the interventional scan (PET/CT) or the conventional scan (standard CT) to look for a source of infection. Diagnostic yield, change in management and outcomes will be compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* About to have an allogeneic haematopoietic stem cell transplant, OR
* About to have an autologous haematopoietic stem cell transplant, OR
* Commencing induction or consolidation chemotherapy with curative intent for acute myeloid or acute lymphoid leukaemia

Exclusion Criteria:

* Current actively diagnosed infection prior to transplant or chemotherapy
* Allergy to intravenous contrast for CT imaging
* eGFR <30
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Change in management following randomized scan | Within 48 hours of scan result
  Defined as:
  * referral for targeted sampling, referral for surgery
  * change in antimicrobial therapy
  * removal of a central line

SECONDARY OUTCOMES:
Proportion of participants with a cause of neutropenic fever | By hospital discharge, an average of 4 weeks
  The proportion of participants in each arm where there is a confirmed cause of neutropenic fever
Hospital length of stay | By hospital discharge, an average of 4 weeks
  The duration (in days) of hospital length of stay for the episode in which neutropenic fever occurred
Costs of hospital care | By hospital discharge, an average of 4 weeks
  The overall cost of the inpatient stay for the episode in which neutropenic fever occurred
Proportion admitted to intensive care | By hospital discharge, an average of 4 weeks
  The proportion of patients in each arm who were admitted to intensive care during their admission in which neutropenic fever occurred
In hospital mortality | By hospital discharge, an average of 4 weeks
  The proportion of patients per arm who have passed away during the admission in which neutropenic fever occurred
6 month mortality | 6 months from study entry
  The proportion of patients per arm who have passed away 6 months post study entry

CONTACTS AND LOCATIONS:
Overall Officials: Monica Slavin, MBBS, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Melbourne Health, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tew M, Douglas AP, Szer J, Bajel A, Harrison SJ, Tio SY, Worth LJ, Hicks RJ, Ritchie D, Slavin MA, Thursky KA, Dalziel K. Evaluating the cost-effectiveness of [18F]FDG-PET/CT for investigation of persistent or recurrent neutropenic fever in high-risk haematology patients. Cancer Imaging. 2023 Dec 15;23(1):119. doi: 10.1186/s40644-023-00647-7. PMID 38102639
- [Derived] Douglas A, Thursky K, Spelman T, Szer J, Bajel A, Harrison S, Tio SY, Bupha-Intr O, Tew M, Worth L, Teh B, Chee L, Ng A, Carney D, Khot A, Haeusler G, Yong M, Trubiano J, Chen S, Hicks R, Ritchie D, Slavin M. [18F]FDG-PET-CT compared with CT for persistent or recurrent neutropenic fever in high-risk patients (PIPPIN): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Haematol. 2022 Aug;9(8):e573-e584. doi: 10.1016/S2352-3026(22)00166-1. Epub 2022 Jun 28. PMID 35777413